CLINICAL TRIAL: NCT02913534
Title: Hypofractionated Stereotactic Radiation Therapy of Brain Metastases: Evaluation of Whole-brain Radiotherapy
Status: Completed | Type: Observational
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Other Study IDs: ICL_2014_0001
Record Dates: First submitted 2016-09-22; First posted 2016-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Brain Metastasis
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

INTERVENTIONS:
Radiation: whole brain radiotherapy

SUMMARY:
The aim is to identify in patients with brain metastases the predictive factors of overall survival, survival without local recurrence and survival with progression-free brain metastases after complementary whole brain radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one to three brain metastases treated in our department with hypofractionated stereotactic radiotherapy (SRT) from March 2008 to February 2013.

Exclusion Criteria:

* A patient record captured after February 2013.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients records would be extracted from the electronic health record system of Institut de Cancérologie de Lorraine.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Overall survival | 72 months

CONTACTS AND LOCATIONS:
Overall Officials: PHILIPPE ROYER, MD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy, France